CLINICAL TRIAL: NCT04839887
Title: Factors Affecting the Quality of Life After Ischemic Stroke in Young Adults: a Prospective Observational Study in Young Ischemic Stroke Patients Under 50 Years
Brief Title: Factors Affecting the Quality of Life After Ischemic Stroke in Young Adults
Acronym: FRAILTY
Status: Recruiting | Type: Observational
Sponsor: Elena Gurkova (Other)
Collaborators: University Hospital Olomouc (Other)
Responsible Party: Sponsor-Investigator, Elena Gurkova, Associated professor, Palacky University
Organization: Palacky University (Other)
Other Study IDs: NU21-09-00053
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke
Keywords: Young Ischemic Stroke; Stroke recovery; Health-Related Quality of Life; Life Change Events; Life Experiences
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Validation study: Three hundred patients with ischemic stroke (18-65 years) will be enrolled for the validation of the Czech version of the the Stroke Impact Scale 3.0. The reliability and validity study will have a cross-sectional design.
- Prospective quantitative study: Two hundred enrolled IS patients (100 young IS patients < 50 years and 100 IS patients of 50-65 years) will undergo a serial of structured and standardized questionnaires during scheduled outpatients' controls three, six and 12 months after IS. In all enrolled patients, the functional outcome, neuropsychological status and quality of life will be assessed using standardized scales and tools.
- In-depth interview qualitative study: twenty young IS patients < 50 years will undergo an in-depth, semi-structured interview with explanatory questions that will allow a detailed understanding of the patient's experience. Interpretative phenomenological analysis (IPA) study design will be used.

SUMMARY:
Despite a generally favourable 3-month functional outcome and a very low mortality, young ischemic stroke (IS) patients face to reduced quality of life associated with a complexity of problems or "invisible dysfunctions" after IS. Better identification and understanding to these factors may improve stroke rehabilitation and stroke self-management programmes, wich will lead to better stroke recovery. The aim of the study is to assess the predictors of the health-related quality of life in young patients under 50 years after ischemic stroke, and to to evaluate specific changes in different dimensions of health-related quality of life during the first year of post-stroke recovery using a standardized battery of neuropsychological tools and stroke specific health-related quality of life measures. In the first phase of the study, 300 IS patients will be enrolled for the validation of the Czech version of the the Stroke Impact Scale 3.0. In the second phase of study, 200 enrolled IS patients (100 young IS patients < 50 years and 100 IS patients of 50-65 years) will undergo a serial of structured and standardized questionnaires during scheduled outpatients' controls three, six and 12 months after IS. In the third phase of study, twenty young IS patients < 50 years will undergo an in-depth, semi-structured interview with explanatory questions that will allow a detailed understanding of the patient's experience. Interpretative phenomenological analysis (IPA) study design will be used.

DETAILED DESCRIPTION:
Despite a generally favourable 3-month functional outcome and a very low mortality, young ischemic stroke (IS) patients face to reduced quality of life associated with a complexity of problems or "invisible dysfunctions" after IS. Fatigue, cognitive impairment, anxiety, depression, sexual dysfunction, loss of employment, social isolation, lack of specialist support, reduction in mobility and life roles, negative body image, impaired self-efficacy and self-esteem are considered most relevant factors. Investigation of predictors of post-stroke quality of life in young-onset patients is needed to design, implement, and evaluate specific young stroke rehabilitation and stroke self-management programmes.

The aim of the study is to assess the predictors of the health-related quality of life in young patients under 50 years after ischemic stroke, and to evaluate specific changes in different dimensions of health-related quality of life during the first year of post-stroke recovery using a standardized battery of neuropsychological tools and stroke specific health-related quality of life measures. The aims of the study will be met by the triangulation of qualitative and quantitative research methods.

In the first phase of the study, 300 IS patients will be enrolled for the validation of the Czech version of the the Stroke Impact Scale 3.0. The reliability and validity study will have a cross-sectional design. In the second phase of study, 200 enrolled IS patients (100 young IS patients < 50 years and 100 IS patients of 50-65 years) will undergo a serial of structured and standardized questionnaires during scheduled outpatients' controls three, six and 12 months after IS. In all enrolled patients, the functional outcome, neuropsychological status and quality of life will be assessed using standardized scales and tools. In the third phase of study, twenty young IS patients < 50 years will undergo an in-depth, semi-structured interview with explanatory questions that will allow a detailed understanding of the patient's experience. Interpretative phenomenological analysis (IPA) study design will be used.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Age 18-65 years

Exclusion Criteria:

* Transient ischemic attack without progression to ischemic stroke
* Haemorrhagic stroke
* Severe cognitive impairment
* Severe communication disorder (sensory aphasia with the inability to understand having been verified by a certified speech therapist)
* Concomitant severe systemic illness
* Impaired ability to understand the questionnaires

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from individuals, diagnosed with ischemic stroke according to the ICD-10 classification who will be admitted to the stroke unit.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Stroke Impact Scale (version 3.0) | three, six and 12 months after stroke
  Assessment of the impact of stroke on eight domains relating to self-rated quality of life, self-perceived disability, and global recovery after stroke (i.e., strength, hand function, mobility, physical and instrumental activities of daily living, memory and thinking, communication, emotion, and social participation). Scores for each domain range from 0 to 100, and higher scores indicate a better health related quality of life

SECONDARY OUTCOMES:
Change of the World Health Organization Quality of Life - BREF version (WHOQOL-BREF, self-reported) | three, six and 12 months after stroke
  Assessment of four domains relating to quality of life (Physical health, Psychological domain, Social relationships, Environment). The four domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. The domain scores will be transformed in accordance with two transformation methods outlined in the WHOQOL-BREF scoring instructions. The domain scores will be transformed into scores ranging between 4 and 20 points (the first transformation method) or into a linear scale between 0 and 100 points (the second transformation method)
Change of the Barthel Index of Activities of Daily Living (self-reported) | three, six and 12 months after stroke
  Measure of performance in activities of daily living. Measure of performance in activities of daily living. Scores of 10 personal activities range from 0 to 100 points and higher score indicates greater independence.
Change of Modified Rankin Scale (self-reported) | three, six and 12 months after stroke
  Scale used for measuring the degree of disability or dependence in the daily activities in patients after stroke. Most widely used clinical outcome measure after stroke. Scale has six points and higher score means worse outcome; minimum is 0 points indicating no symptoms at all and maximum is 6 points indicating death.
Change of post-stroke depression and anxiety (self-reported) | three, six and 12 months after stroke
  Assessment of depressive and anxiety symptoms using Beck Depression Inventory II and Hospital Anxiety and Depression Scale. Higher total scores indicate more severe depressive symptoms.
Change of the Montreal Cognitive Assessment (MoCA) | three, six and 12 months after stroke
  Assessment of cognitive functions (cognitive test measuring specific cognitive domains). The MoCA generates a total score and six domain-specific index scores: Memory, Executive Functioning, Attention, Language, Visuospatial, and Orientation. MoCA score range between 0 and 30. Higher score indicates better cognitive functions. The following ranges are used to grade the severity of cognitive impairment: 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment.
Change from 3-month the lived experience of ischemic stroke of young patients up to 50 years at 12 months. | three and 12 months after stroke
  Semi-structured interviews with stroke patients
Change in the NIH Stroke Scale (NIHSS) | three, six and 12 months after stroke
  NIHSS is used to objectively quantify the impairment caused by a stroke. Higher score indicates more severe neurological deficit.

OTHER OUTCOMES:
Change in the Fatigue Severity Scale | three, six and 12 months after stroke
  Assessment of post-stroke fatigue using Fatigue Severity Scale. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. The minimum score is nine and the highest is 63 points. The higher score indicates more severe fatigue and greater affecting of the person's activities.
Change in the Brief Pain Inventory | three, six and 12 months after stroke
  Includes questions on site of pain, severity of pain, and how pain interfered with the patient's mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. These questions are rated on a scale of 0 to 10; a higher score indicates greater pain or greater interference with the daily activities.
Change in the Multi-dimensional Scale of Perceived Social Support | three, six and 12 months after stroke
  The Multi-dimensional Scale of Perceived Social Support (MSPSS) assesses different sources of support. The MSPSS is a brief 12-item, self-administered measurement tool with three subscales: Family, Friends, and Significant Others. A higher score indicates greater social support perceived by an individual; the total possible score ranges between 12 and 84 points.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Gurkova, PhD, Principal Investigator — Palacky University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Palacky University, Faculty of Health Sciences, Olomouc, Czechia

REFERENCES:
- [Result] Arntz RM, van Alebeek ME, Synhaeve NE, Brouwers PJ, van Dijk GW, Gons RA, den Heijer T, de Kort PL, de Laat KF, van Norden AG, Vermeer SE, van der Vlugt MJ, Kessels RP, van Dijk EJ, de Leeuw FE. Observational Dutch Young Symptomatic StrokE studY (ODYSSEY): study rationale and protocol of a multicentre prospective cohort study. BMC Neurol. 2014 Mar 22;14:55. doi: 10.1186/1471-2377-14-55. PMID 24655479
- [Result] Bartholome L, Winter Y. Quality of Life and Resilience of Patients With Juvenile Stroke: A Systematic Review. J Stroke Cerebrovasc Dis. 2020 Oct;29(10):105129. doi: 10.1016/j.jstrokecerebrovasdis.2020.105129. Epub 2020 Jul 15. PMID 32912563
- [Result] Boot E, Ekker MS, Putaala J, Kittner S, De Leeuw FE, Tuladhar AM. Ischaemic stroke in young adults: a global perspective. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):411-417. doi: 10.1136/jnnp-2019-322424. Epub 2020 Feb 3. PMID 32015089
- [Result] de Bruijn MA, Synhaeve NE, van Rijsbergen MW, de Leeuw FE, Mark RE, Jansen BP, de Kort PL. Quality of Life after Young Ischemic Stroke of Mild Severity Is Mainly Influenced by Psychological Factors. J Stroke Cerebrovasc Dis. 2015 Oct;24(10):2183-8. doi: 10.1016/j.jstrokecerebrovasdis.2015.04.040. Epub 2015 Jul 26. PMID 26215135
- [Result] Douven E, Schievink SH, Verhey FR, van Oostenbrugge RJ, Aalten P, Staals J, Kohler S. The Cognition and Affect after Stroke - a Prospective Evaluation of Risks (CASPER) study: rationale and design. BMC Neurol. 2016 May 12;16:65. doi: 10.1186/s12883-016-0588-1. PMID 27176617
- [Result] Ekker MS, Boot EM, Singhal AB, Tan KS, Debette S, Tuladhar AM, de Leeuw FE. Epidemiology, aetiology, and management of ischaemic stroke in young adults. Lancet Neurol. 2018 Sep;17(9):790-801. doi: 10.1016/S1474-4422(18)30233-3. PMID 30129475
- [Result] Harno H, Haapaniemi E, Putaala J, Haanpaa M, Makela JP, Kalso E, Tatlisumak T. Central poststroke pain in young ischemic stroke survivors in the Helsinki Young Stroke Registry. Neurology. 2014 Sep 23;83(13):1147-54. doi: 10.1212/WNL.0000000000000818. Epub 2014 Aug 15. PMID 25128182
- [Result] Heiberg G, Friborg O, Pedersen SG, Thrane G, Holm Stabel H, Feldbaek Nielsen J, Anke A. Post-stroke health-related quality of life at 3 and 12 months and predictors of change in a Danish and Arctic Norwegian Region. J Rehabil Med. 2020 Sep 8;52(9):jrm00096. doi: 10.2340/16501977-2716. PMID 32735024
- [Result] Kapoor A, Scott C, Lanctot KL, Herrmann N, Murray BJ, Thorpe KE, Lien K, Sicard M, Swartz RH. Symptoms of depression and cognitive impairment in young adults after stroke/transient ischemic attack. Psychiatry Res. 2019 Sep;279:361-363. doi: 10.1016/j.psychres.2019.06.022. Epub 2019 Jul 1. PMID 31272664
- [Result] Kono Y, Terasawa Y, Sakai K, Iguchi Y, Nishiyama Y, Nito C, Suda S, Kimura K, Kanzawa T, Imafuku I, Nakayama T, Ueda M, Iwanaga T, Kono T, Yamashiro K, Tanaka R, Okubo S, Nakajima M, Nakajima N, Mishina M, Yaguchi H, Oka H, Suzuki M, Osaki M, Kaneko N, Kitagawa K, Okamoto S, Nomura K, Yamazaki M, Nagao T, Murakami Y. Risk factors, etiology, and outcome of ischemic stroke in young adults: A Japanese multicenter prospective study. J Neurol Sci. 2020 Oct 15;417:117068. doi: 10.1016/j.jns.2020.117068. Epub 2020 Jul 29. PMID 32745720
- [Result] Lam KH, Blom E, Kwa VIH. Predictors of quality of life 1 year after minor stroke or TIA: a prospective single-centre cohort study. BMJ Open. 2019 Nov 2;9(11):e029697. doi: 10.1136/bmjopen-2019-029697. PMID 31678939
- [Result] Maaijwee NA, Arntz RM, Rutten-Jacobs LC, Schaapsmeerders P, Schoonderwaldt HC, van Dijk EJ, de Leeuw FE. Post-stroke fatigue and its association with poor functional outcome after stroke in young adults. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1120-6. doi: 10.1136/jnnp-2014-308784. Epub 2014 Oct 31. PMID 25362090
- [Result] McKevitt C, Redfern J, Mold F, Wolfe C. Qualitative studies of stroke: a systematic review. Stroke. 2004 Jun;35(6):1499-505. doi: 10.1161/01.STR.0000127532.64840.36. Epub 2004 Apr 22. PMID 15105517
- [Result] Pinter D, Enzinger C, Gattringer T, Eppinger S, Niederkorn K, Horner S, Fandler S, Kneihsl M, Krenn K, Bachmaier G, Fazekas F. Prevalence and short-term changes of cognitive dysfunction in young ischaemic stroke patients. Eur J Neurol. 2019 May;26(5):727-732. doi: 10.1111/ene.13879. Epub 2019 Jan 9. PMID 30489673
- [Result] Rhudy LM, Wells-Pittman J, Flemming KD. Psychosocial Sequelae of Stroke in Working-Age Adults: A Pilot Study. J Neurosci Nurs. 2020 Aug;52(4):192-199. doi: 10.1097/JNN.0000000000000523. PMID 32511173
- [Result] Schneider S, Taba N, Saapar M, Vibo R, Korv J. Determinants of Long-Term Health-Related Quality of Life in Young Ischemic Stroke Patients. J Stroke Cerebrovasc Dis. 2021 Feb;30(2):105499. doi: 10.1016/j.jstrokecerebrovasdis.2020.105499. Epub 2020 Nov 30. PMID 33271487
- [Result] Synhaeve NE, Arntz RM, Maaijwee NA, Rutten-Jacobs LC, Schoonderwaldt HC, Dorresteijn LD, de Kort PL, van Dijk EJ, de Leeuw FE. Poor long-term functional outcome after stroke among adults aged 18 to 50 years: Follow-Up of Transient Ischemic Attack and Stroke Patients and Unelucidated Risk Factor Evaluation (FUTURE) study. Stroke. 2014 Apr;45(4):1157-60. doi: 10.1161/STROKEAHA.113.004411. Epub 2014 Feb 27. PMID 24578210
- [Result] Rutten-Jacobs LC, Maaijwee NA, Arntz RM, Van Alebeek ME, Schaapsmeerders P, Schoonderwaldt HC, Dorresteijn LD, Overeem S, Drost G, Janssen MC, van Heerde WL, Kessels RP, Zwiers MP, Norris DG, van der Vlugt MJ, van Dijk EJ, de Leeuw FE. Risk factors and prognosis of young stroke. The FUTURE study: a prospective cohort study. Study rationale and protocol. BMC Neurol. 2011 Sep 20;11:109. doi: 10.1186/1471-2377-11-109. PMID 21933424
- [Result] Zawawi NSM, Aziz NA, Fisher R, Ahmad K, Walker MF. The Unmet Needs of Stroke Survivors and Stroke Caregivers: A Systematic Narrative Review. J Stroke Cerebrovasc Dis. 2020 Aug;29(8):104875. doi: 10.1016/j.jstrokecerebrovasdis.2020.104875. Epub 2020 May 23. PMID 32689648
- [Derived] Sanakova S, Gurkova E, Bartonickova D, Sturekova L, Franc D, Zapletalova J, Divisova P, Sanak D. Post-Stroke Fatigue in Patients at 3 Months After Ischemic Stroke: Analysis From the FRAILTY Study. SAGE Open Nurs. 2025 Nov 26;11:23779608251400226. doi: 10.1177/23779608251400226. eCollection 2025 Jan-Dec. PMID 41321434
- [Derived] Sanakova S, Gurkova E, Sturekova L, Bartonickova D, Machalkova L, Mazalova L. How to return? experiences of patients in working age after first Ischaemic stroke: an interpretative phenomenological analysis of patient s perspective at 12 - 24 months post-stroke. Int J Qual Stud Health Well-being. 2024 Dec;19(1):2398249. doi: 10.1080/17482631.2024.2398249. Epub 2024 Sep 4. PMID 39229807
- [Derived] Sanak D, Gurkova E, Sturekova L, Sanakova S, Zapletalova J, Franc D, Bartonickova D. Quality of Life in Patients with Excellent 3-Month Clinical Outcome after First-Ever Ischemic Stroke: A Time to Redefine Excellent Outcome? Eur Neurol. 2024;87(1):1-10. doi: 10.1159/000535685. Epub 2024 Jan 17. PMID 38232714